CLINICAL TRIAL: NCT07266805
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, 3-Part Study to Evaluate the Efficacy and Safety of Orally Administered Deucrictibant Extended-release (XR) Tablet for Prophylaxis and Deucrictibant Immediate-release (IR) Capsule for On-demand Treatment of Angioedema Attacks in Adults With Acquired Angioedema Due to C1 Inhibitor Deficiency
Brief Title: Study of Oral Deucrictibant XR Tablet for Prophylaxis and Deucrictibant IR Capsule for On-Demand Treatment of Angioedema Attacks in Adults With Acquired Angioedema Due to C1 Inhibitor Deficiency
Acronym: CREAATE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pharvaris Netherlands B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PHA022121-C308
Record Dates: First submitted 2025-10-20; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acquired Angioedema Due to C1-Inhibitor Deficiency (AAE-C1-INH)
Keywords: Acquired Angioedema-C1-INH; AAE-C1-INH; Oral Treatment; deucrictibant; Prophylaxis; On-demand; C1-Inhibitor Deficiency; PHA121; Pharvaris; Bradykinin B2 Receptor Antagonists; Angioedema; Acquired; Acquired angioedema
MeSH Terms: conditions — Angioedemas, Hereditary; Angioedema; Acquired angioedema

STUDY DESIGN:
Intervention Model Description: Part 1 is parallel Part 2 is crossover Part 3 is single group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1 - Arm 1 - Active (Experimental)
  Interventions: Drug: Deucrictibant
- Part 1 - Arm 2 - Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2 - Arm 1 (Experimental)
  Interventions: Drug: Deucrictibant; Drug: Placebo
- Part 2 - Arm 2 (Experimental)
  Interventions: Drug: Deucrictibant; Drug: Placebo
- Part 3 - Open-label (Experimental)
  Interventions: Drug: Deucrictibant

INTERVENTIONS:
Drug: Deucrictibant — Part 1: Deucrictibant 40 mg extended-release tablet for once daily oral use
  Arms: Part 1 - Arm 1 - Active
Drug: Placebo — Part 1: Placebo Comparator tablet for once daily oral use
  Arms: Part 1 - Arm 2 - Placebo
Drug: Deucrictibant — Part 2: Deucrictibant 20 mg soft capsule oral use
  Arms: Part 2 - Arm 1; Part 2 - Arm 2
Drug: Placebo — Part 2: Placebo Comparator soft capsule oral use
  Arms: Part 2 - Arm 1; Part 2 - Arm 2
Drug: Deucrictibant — Part 3: Deucrictibant 20 mg soft capsule oral use
  Arms: Part 3 - Open-label

SUMMARY:
This is a Phase 3, multicenter, 3-part study, with 2 randomized, double-blind, placebo-controlled parts and an open-label extension part, to evaluate the efficacy and safety of orally administered deucrictibant XR tablet for prophylaxis, and deucrictibant IR capsule for on-demand treatment of angioedema attacks in adult participants aged ≥ 18 years with AAE-C1INH.

DETAILED DESCRIPTION:
The study consists of a Screening Period, during which eligibility is confirmed, a Part 1 Prophylaxis Double-blind Treatment Phase, a Part 2 On-demand, Double-blind Treatment Phase, and a Part 3 On-demand Open-label Extension Phase. Approximately 24 participants will be randomized in Part 1 into 2 parallel arms for a treatment period of 12 weeks. During the prophylaxis treatment period participants will receive blinded study drug (deucrictibant 40 mg XR or placebo randomized in a 1:1 ratio). Upon completion of Part 1, participants will roll-over into Part 2. In addition to rollover participants completing Part 1, new deucrictibant treatment-naïve participants will be enrolled directly into Part 2 and this may occur while Part 1 is ongoing. During the on-demand period participants will receive blinded study drug (deucrictibant 20 mg IR capsule or matching placebo randomized in a 1:1 ratio, 2-period, 2-treatment crossover design) for 2 qualifying AAE-C1INH attacks. Participants completing Part 2 may roll over into Part 3 where all AAE-C1INH attacks will be treated with open-label deucrictibant 20 mg soft capsule.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Male or female (sex at birth) aged ≥18 years
* Diagnosis of AAE-C1INH
* History of AAE-C1INH attacks prior to the Screening Visit:
* Participants enrolling in Part 1 must have stable underlying disease of AAE-C1INH

  * The underlying condition can reasonably be expected to remain stable for the duration
* Reliable access and ability to use available therapy to effectively manage AAE- C1INH attacks.
* Female participants of childbearing potential must agree to the protocol-specified pregnancy testing and to be abstinent from heterosexual intercourse or to use an acceptable contraception method.

Females of non-childbearing potential (prepubertal, surgically sterile, or postmenopausal with ≥ 12 months amenorrhea and postmenopausal FSH confirmation) are not required to use contraception during the study.

• Capable of recording, without assistance, eDiary and ePRO data using an electronic device, as evidenced by the eDiary and ePRO training.

Exclusion Criteria:

* Participation in a clinical study with any other investigational drug within the last 30 days or within 5 half-lives of the investigational drug at the Screening Visit (whichever is longer).
* Participants who have previously received prophylactic therapy but have stopped can participate in this study provided the last dose of the treatment was received prior to the timepoint before the Screening Visit
* Any females who are pregnant, plan to become pregnant, or are currently breast-feeding
* Abnormal hepatic function
* Moderate or severe renal impairment
* Any clinically significant comorbidity or systemic dysfunction that would interfere with the participant's safety or ability to participate in the study.
* History of epilepsy and/or other significant neurological diseases
* Any clinically significant and uncontrolled gastrointestinal dysfunction that may impact study drug absorption
* Evidence of current alcohol or drug abuse
* Use of medications that are moderate and strong inhibitors of cytochrome P450 (CYP) 3A4, or strong inducers of CYP3A4 within the last 30 days or within 5 half-lives (whichever is longer) at the time of the Screening Visit
* Known hypersensitivity to deucrictibant or any of the excipients of the study drug
* Use of angiotensin-converting enzyme inhibitors or any estrogen-containing medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Time-normalized number of Investigator-confirmed AAE attacks during Treatment Phase
Part 2 (On-demand, Double-blind Treatment Phase) | 12 hours post-treatment
  Time to symptom relief, Patient Global Impression of Change (PGI-C) rating of at least "better"
Part 3 (On-demand, Open-label Extension Treatment Phase) | Through study completion, an average of 36 weeks
  Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and TEAEs leading to study drug discontinuation

SECONDARY OUTCOMES:
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Proportion of participants who are AAE attack-free during Treatment Phase
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Time-normalized number of Investigator-confirmed AAE attacks treated with on-demand medication during Treatment Phase
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Time-normalized number of Investigator-confirmed moderate or severe AAE attacks during Treatment Phase
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Safety endpoints: Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and TEAEs leading to study drug discontinuation
Part 1 (Prophylaxis, Double-blind Treatment Phase) | 12 weeks
  Pharmacokinetics [PK]: Deucrictibant singular plasma concentration
Part 1 (Prophylaxis, Double-blind Treatment Phase) | From enrollment through end of Part 1 (Week 12)
  Patient reported outcomes:
  · Patient reported outcome: Angioedema Quality of Life (AE-QoL) questionnaire
  The AE-QoL is a short 17-item questionnaire designed to retrospectively assess HRQoL, with a recall period of 4 weeks. Its results can be displayed as a total score or as 4 domain scores. The scores range from 0 to 100, after linear transformation of raw values, with higher scores indicating higher HRQoL impairment.
Part 1 (Prophylaxis, Double-blind Treatment Phase) | From enrollment through end of Part 1 (Week 12)
  Patient reported outcomes:
  · Patient Global Assessment of Change (PGA-Change)
  PGA-Change assesses on a 5-point scale how the participant's QoL has been impacted by HAE since start taking the study drug
Part 1 (Prophylaxis, Double-blind Treatment Phase) | From enrollment through end of Part 1 (Week 12)
  Patient reported outcomes:
  · Angioedema Control Test 4-week version (AECT-4wk)
  AECT-4wk measures disease control retrospectively, it comprises 4 questions over a 4-week recall period. Scores for the responses in the AECT range from 0 to 16, with higher scores indicating better disease control (≤ 9 poorly controlled; ≥ 10 well controlled)
Part 1 (Prophylaxis, Double-blind Treatment Phase) | From enrollment through end of Part 1 (Week 12)
  Patient reported outcomes:
  · EuroQol 5 Dimension 5 level (EQ 5D 5L)
  EQ 5D 5L is a brief, multiattribute, generic, health status measure composed of 5 questions with Likert response options (descriptive system) and a visual analog scale (EQ-VAS). The latter asks patients to rate their own health from 0 to 100 (the worst and best imaginable health, respectively)
Part 2 (On-demand, Double-blind Treatment Phase) | 48 hours post-treatment
  Time to complete symptom resolution, Patient Global Impression of Severity (PGI-S) rating of "no symptoms
Part 2 (On-demand, Double-blind Treatment Phase) | 12 hours post-treatment
  Time to symptom relief defined as PGI-S rating of at least 1 point reduction
Part 2 (On-demand, Double-blind Treatment Phase) | 12 weeks
  Safety endpoints: Incidence of treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), and TEAEs leading to study drug discontinuation
Part 2 (On-demand, Double-blind Treatment Phase) | Day 1
  Pharmacokinetics [PK]: Deucrictibant plasma concentration-time profiles

OTHER OUTCOMES:
Part 3 (On-demand, Open-label Extension Treatment Phase) | 12 hours post-treatment
  Time to symptom relief, as PGI-C rating of at least "better"

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Pharvaris, Study Director — Pharvaris Netherlands B.V.
Locations (2):
- United States (2):
  - Study Site, Walnut Creek, California
  - Study Site, St Louis, Missouri